CLINICAL TRIAL: NCT01496638
Title: How Should Coronary Artery Stenoses With Significant Side Branch be Stented? A Strategy of Stenting Both Main Vessel and Side Branch Compared to a Strategy of Stenting the Main Vessel and Only Stenting the Side Branch if Necessary.
Brief Title: The Nordic-Baltic Bifurcation Study IV
Acronym: BIF IV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Evald Hoej Christiansen (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor-Investigator, Evald Hoej Christiansen, MD, Aarhus University Hospital Skejby
Organization: Aarhus University Hospital Skejby (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20080192
Record Dates: First submitted 2011-12-19; First posted 2011-12-21 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
Keywords: PCI; Bifurcation lesion
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- "No side branch treatment" group (Experimental): Implantation of coronary stent in bifurcation lesion
  Interventions: Procedure: Implantation of coronary stent in bifurcation lesion
- "Stenting of main vessel and side branch" group (Experimental): Implantation of coronary stent in bifurcation lesion
  Interventions: Procedure: Implantation of coronary stent in bifurcation lesion

INTERVENTIONS:
Procedure: Implantation of coronary stent in bifurcation lesion — Implantation of coronary stent in bifurcation lesion with no side branch treatment
  Other Names: PCI; PTCA
  Arms: "No side branch treatment" group
Procedure: Implantation of coronary stent in bifurcation lesion — Implantation of coronary stent in bifurcation lesion with stenting of main vessel and side branch
  Other Names: PCI; PTCA
  Arms: "Stenting of main vessel and side branch" group

SUMMARY:
How should coronary artery stenoses with significant side branch be stented?

A strategy of stenting both main vessel and side branch compared to a strategy of stenting the main vessel and only stenting the side branch if necessary.

The 2-stent strategy is superior to the 1-stent strategy regarding occurrence of cardiac death, non-procedure related myocardial infarction and re-revascularization with percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG).

DETAILED DESCRIPTION:
Design:

* Randomised open multicentre trial.

Patients:

* Number 450.

Randomisation:

* No side branch treatment group or stenting of main vessel and side branch group.

Evaluation of endpoints:

* Primary and secondary endpoints will be assessed by an independent endpoint committee.
* The endpoint committee will consist of experienced cardiologists with professor Kristian Thygesen, Aarhus Universitetshospital, as chairman.

Sample size calculation:

* A total of 225 patients will be included in each group, in total 450 patients. We expect a primary endpoint rate of 10% (cardiac death, non-procedure related myocardial infarction related to index lesion or TLR after 6 months) in the 1- stent strategy group and of 3% in the 2-stent strategy group. With an alpha of 5% and a strength of 80%, 194 patients will be needed in each group (two-sided chi-square test) to demonstrate this difference. The expected primary endpoint rate after 6 months is based on 6 months MACE rates and on the angiographic results in our previously published studies. In these studies, a 6 months MACE rate of 3.7% was found in the culotte group of the Nordic Stent Technique Study. Besides, an angiographic restenosis rate of 19.2% in the 1-stent strategy group in the Nordic Bifurcation Study is estimated to translate to a MACE rate of approximately 10% in the present study.

Analysis of the population:

* The results will be analyzed according to the intention-to-treat principle.

Data management:

* The study is reported to Datatilsynet (The Danish Data Protection Agency) and the agency's guidelines for data management will be followed.

Dedicated case record forms (CRF) will be used and faxed to PCI research, Cardiac Cath. Lab., Aarhus University Hospital, Skejby, DK-8200 Aarhus N, Denmark. Data will be stored in an Access database and double data entry will be used as quality control. There will be a log of accesses and attempt of accesses. Back-up data and original data will be cryptotized.

Monitoring of the study:

* The study will be monitored according to the GCP rules by independent professionals. During the study period, monitors will have regular contact to the participating departments to ensure that the trial is conducted in compliance with the protocol, GCP and applicable regulatory requirements

Publication:

* Results, positive as well as negative, will be published in an international cardiovascular journal. Publication and author issues will be decided by the steering committee on basis of general involvement in the study (drafting of protocol, core lab. function, end point committee membership, etc.) and of number of included patients.

ELIGIBILITY:
Inclusion Criteria:

* Stable or unstable angina pectoris or silent angina pectoris.
* Genuine bifurcation lesion ( Medina type 1,1,1 or 1,0,1 or 0,1,1)
* Lesion of "LAD/diagonal", "Cx/obtuse marginal", "RCA-PDA/posterolateral branch" or "LM/Cx/LAD".
* Diameter of main vessel by visual estimate >3.0 mm.
* Diameter of side branch by visual estimate >2.75 mm.
* Signed informed consent.

Exclusion Criteria:

* ST-elevation infarction within 24 hours.
* Side branch lesion length >15 mm.
* Expected survival < 1 year.
* S-creatinine >200 µmol/l.
* Allergy to Aspirin, Clopidogrel or Ticlopidine.
* Allergy to Sirolimus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Combined endpoint of: Cardiac death, non-index procedure related myocardial infarction or target lesion revascularisation | After 6 months

SECONDARY OUTCOMES:
MACE (cardiac death, non-index procedure related myocardial infarction, stent thrombosis or target lesion revasculation) | During admission, after 1, 24, 36 and 60 months.
Cardiac death. | During the admission, after 1, 6, 24, 36 and 60 months.
Non-index procedure related myocardial infarction during the admission. | After 1, 6, 24, 36 and 60 months.
Stent thrombosis. | During admission, after 1, 6, 24, 36 and 60 months.
Total mortality | During admission, after 1, 6, 24, 36 and 60 months and 10 years.
target lesion revascularisation. | During admission, after 1, 6, 24, 36 and 60 months.
target vessel revascularisation. | During admission, after 1, 6, 24, 36 and 60 months.
Index procedure related myocardial infarction based on biomarkers (CK-MB mass, TNT/TNI | During hospital period, 1, 8, 24, 36 and 60 months
CCS angina class | After 6, 8, 24, 36 and 60 months.

CONTACTS AND LOCATIONS:
Overall Officials: Niels R Holm, MD, Principal Investigator — MD
Locations (1):
- Aarhus University Hospital, Skejby, Aarhus N, Denmark

REFERENCES:
- [Derived] Kumsars I, Holm NR, Niemela M, Erglis A, Kervinen K, Christiansen EH, Maeng M, Dombrovskis A, Abraitis V, Kibarskis A, Trovik T, Latkovskis G, Sondore D, Narbute I, Terkelsen CJ, Eskola M, Romppanen H, Laine M, Jensen LO, Pietila M, Gunnes P, Hebsgaard L, Frobert O, Calais F, Hartikainen J, Aaroe J, Ravkilde J, Engstrom T, Steigen TK, Thuesen L, Lassen JF; Nordic Baltic bifurcation study group. Randomised comparison of provisional side branch stenting versus a two-stent strategy for treatment of true coronary bifurcation lesions involving a large side branch: the Nordic-Baltic Bifurcation Study IV. Open Heart. 2020 Jan 19;7(1):e000947. doi: 10.1136/openhrt-2018-000947. eCollection 2020. PMID 32076558